CLINICAL TRIAL: NCT01302782
Title: The Effects of Normobaric Hypoxia on Blood Glucose Levels.
Status: Withdrawn | Type: Observational
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FWH20110021H
Record Dates: First submitted 2011-02-17; First posted 2011-02-24 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Glucose
Keywords: Altitude; Glucose

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to observe whether there is a change in blood glucose levels in response to a 2 hour oral glucose tolerance tests (OGTT) during acute normobaric hypoxia (short term low oxygen levels at normal ambient air pressure).

ELIGIBILITY:
Inclusion Criteria (non-diabetics):

* Tricare Insurance Beneficiary (military insurance) receiving care at Nellis AFB
* 5 males with a BMI < 25; 5 males with a BMI > 25 at least 18 years of age (MOFH personnel and DoD beneficiaries).
* 5 females with a BMI < 25; 5 females with a BMI > 25 at least 18 years of age (MOFH personnel and DoD beneficiaries).

Exclusion Criteria (non-diabetics):

* History of abnormal fasting glucose.
* Pulmonary disease.
* Any medications that change glucose control to include systemic steroid and diabetic medications.
* History of claustrophobia.
* Pregnant or breast feeding.
* Non-English speaking.
* Physical inability to wear/use the ROBD2

Inclusion Criteria (diabetics):

-5 males and/or females, at least 18 years of age, that are type 2 diabetics (MOFH personnel and DoD beneficiaries).

Exclusion Criteria (diabetics):

* Pulmonary disease.
* History of claustrophobia.
* Pregnant or breast feeding.
* Non-English speaking.
* Physical inability to wear/use the ROBD2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We are recruiting male and female patients (MOFH personnel and DoD beneficiaries) whom are at least 18 years of age from the Nellis Air Force Base population.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in glucose levels at altitude | 1 year
  Subjects will be placed on a Reduced Oxygen Breathing Device (ROBD2) to simulate 3 different altitudes at three separate and distinct time periods (ground, 8,000 feet and 12,000 feet) then obtain c-peptide and 2-hour OGTT to determine blood glucose changes during acute normobaric hypoxia.

CONTACTS AND LOCATIONS:
Overall Officials: Travis Russell, M.D., Principal Investigator — Mike O'Callaghan Federal Hospital/Nellis Air Force Base